CLINICAL TRIAL: NCT03330444
Title: Development of a Non-invasive Diagnosis Tool for the Analysis of the Microbiota to Improve Reproductive Outcomes in Infertile Patients.
Brief Title: Development of a Microbiome Non-invasive Diagnosis Tool
Acronym: ERA-niMIC
Status: Completed | Type: Observational
Sponsor: Igenomix (Industry)
Responsible Party: Sponsor
Other Study IDs: IGX1-MIC-CS-17-05
Record Dates: First submitted 2017-10-24; First posted 2017-11-06 (Actual); Last update posted 2020-10-09 (Actual); Status verified 2020-10

CONDITIONS: Infertility of Uterine Origin
Keywords: Endometrial microbiota; Bacterial pathogens; Assisted reproductive techniques; Dysbiosis; Endometrial receptivity; Endometrial diagnosis
MeSH Terms: conditions — Dysbiosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA from endometrial fluid and biopsy to analyze the endometrial microbiome.
  These samples will be completely exhausted during the analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- LD microbiome receptive to the ERA test: Receptive patients by the ERA test with an endometrial microbiota mainly composed of different species of the genus Lactobacillus, determined by NGS sequencing.
  Interventions: Procedure: Endometrial biopsy and endometrial fluid collection
- NLD microbiome receptive to the ERA test: Receptive patients by the ERA test with an endometrial microbiota composed of different pathogenic bacteria such as Streptococcus and Gardnerella, or not dominated by bacteria of the genus Lactobacillus, determined by NGS sequencing.
  Interventions: Procedure: Endometrial biopsy and endometrial fluid collection

INTERVENTIONS:
Procedure: Endometrial biopsy and endometrial fluid collection — On the same day that the EB for ERA is indicated, in day 5 of a HRT cycle with 5 days of progesterone, according to the common clinical practice, a sample of EF will be aspirated immediately prior to EB for ERA. This EF sample will be used for the non-invasive diagnosis of the microbiome, also a small portion of the endometrial tissue obtained for the endometrial receptivity diagnosis by ERA will be used as a control for the study of the endometrial microbiome. Those patients with a receptive endometrium will continue their ART according to the standard clinical protocol. Those patients with non-receptive endometrium will follow the recommendation derived of the ERA test for the election of the day for a second EB sample, in which the collection of EF sample will be repeated. Finally, the receptivity and microbiome results in EF will be correlated with that on the endometrial tissue, and with the reproductive outcomes of these patients after the embryo transfer.

SUMMARY:
Although the endometrium tissue has been traditionally considered free of bacteria, recent studies have documented the presence of an endometrial microbiome. In a pilot study conducted by our research team, the microorganisms present in the endometrium were analysed in samples of endometrial fluid (EF) using next generation sequencing (NGS).Consistent with previously published studies, in normal conditions the endometrium is mainly composed of different species of the genus Lactobacillus. It was further noted that the presence of other pathogenic bacteria such as Streptococcus, and/or Gardnerella may alter the endometrial microbiome and can disrupt the uterine environment, affecting implantation rates and pregnancy success.

This project aims to validate the microbiome found in the endometrium of women of reproductive age and try to corroborate the relationship between the endometrial microbiome and the reproductive outcomes in patients undergoing assisted reproduction treatment (ART). The use of Endometrial Receptivity Analysis (ERA) tool, together with the analysis of the endometrial flora before the embryo transfer will allow to evaluate the impact of the presence of endometrial pathogens on implantation in receptive patients.

Therefore, the focus of this project is the development and clinical validation of a non-invasive diagnosis tool to analyse the microbiota, adding the microbiome study to the ERA analysis.

DETAILED DESCRIPTION:
Embryonic implantation is a critical process to the survival of the species that is relatively inefficient, especially in humans. Key elements are the embryo, the maternal endometrium, and the cross-communication between them using different scientific perspectives. Endometrial receptivity describes the phenotype that allows embryo adhesion and placentation to occur. Due to the need of an accurate and objective molecular diagnostic test for the receptivity status of endometrium, the Endometrial Receptivity Analysis (ERA) was developed. ERA test is a customized expression microarray that identifies the transcriptomic expression profile signature of the personalized window of implantation (WOI). Its clinical usefulness has been demonstrated in patients with implantation failure in whom 25% of them have a displaced WOI becoming pregnant once the embryo transfer is performed at the proper WOI predicted by ERA. However, this procedure requires an endometrial biopsy (EB), which is the major drawback of this diagnosis test, because embryo transfer has to be delayed to the next cycle, and also the possible discomforts caused to the patients. For this reason, a previous pilot study was conducted in order to confirm whether endometrial receptivity can be predicted through non-invasive methods in endometrial fluid (EF) samples. The gene panel of ERA test was interrogated on epithelial and stromal cells from endometrial biopsies and cells isolated from the EF at the single cell level, demonstrating that the major cells on the EF classifies together with the epithelial population.

On the other hand, to try to better understand the mechanisms that connect endometrial receptivity and/or implantation of the embryo with an altered endometrial microbiome, another pilot study was conducted to determine the composition of the endometrial microbiome after the analysis of the bacterial 16S ribosomal RNA by NGS. Interestingly, in patients with receptive endometrium, diagnosed by Endometrial Receptivity Array (ERA) who had endometrial microbiome with pathogens, or not dominated by bacteria of the genus Lactobacillus (NLD) showed significantly lower implantation (23.1% vs 60.7% p = 0.02), pregnancy (33.3% vs 70.6%, p = 0.03), ongoing pregnancy per embryo transfer (13.3% vs 58.8%, p = 0.03), and live birth (6.7% vs 58.8%, p = 0.002) rates than those with a healthy endometrial microbiome dominated by Lactobacillus (LD). Moreover, this relationship was much more significant when pathogenic species found belonged to the genus Gardnerella and Streptococcus. This is in line with other published studies that analyze the impact of endometrial pathogens in IVF treatments, highlighting the importance of the study of bacterial communities for reproductive health.

Given these preliminary results, the present study aims to validate in a larger sample set, the relationship between the imbalance of endometrial microbiome and the decline in reproductive success in patients undergoing ART. To do this, the experimental design will be improved in the following areas: (i) a higher sample size will be analysed to validate the previous results obtained in the previous pilot study on endometrial microbiome, (ii) paired samples from endometrial fluid and endometrial biopsy will be analysed for the microbial profile to study whether there is bacterial variability associated to the sample type, (iii) the endometrial microbiota will be simultaneously assessed with ERA as a supplementary diagnosis for this tool, and (iv) the analysis of the endometrial microbiota will be performed using the most advanced technology on bacterial metagenome sequencing to widen the information of the microorganisms identified in each sample.

ELIGIBILITY:
Inclusion Criteria:

* Patients in In Vitro Fertilization (IVF) / IntraCytoplasmic Sperm Injection (ICSI) or OVODON with indication of ERA, with or without Preimplantation genetic screening (PGS) indication, which receive embryo transfer with frozen blastocyst stage embryos (day 5/day 6) on a hormone replacement therapy (HRT) cycle.
* Maternal Age: ≤40 years (IVF/ICSI patients)
* Maternal Age: ≤50 years (OVODONATION patients)
* Body Mass Index (BMI): 18.5 - 30 kg / m2 (both inclusive)
* Negative serological tests for human immunodeficiency virus (HIV), hepatitis B virus (HBV), hepatitis C virus (HCV), Rapid plasma reagin (RPR) for syphilis
* Women with regular menstrual formula (3-4 / 26- 35 days)
* Sperm concentration: > 2 million spermatozoa/ml

Exclusion Criteria:

* Patients who are Intra-Uterine Device (IUD) carriers in the last 3 months
* Patients who have taken prescribed antibiotics in the last 3 months before the sample collection. (May be accepted those cases where the patient has received previous prophylactic antibiotics to ovarian puncture in the stimulation cycle, according to the standard clinical practice of the centre. The administration of this antibiotic should be at least 1 month before the sample collection).
* Adnexal or uterine pathologies as uterine malformations that may affect the implantation rate (e.g: Polyps, intramural myoma ≥ 4cm or submucosal, septum, hydrosalpinx, etc). Patients affected (before or after of their inclusion) with any of the previously described pathologies, will be allowed to participate in this study as long as they are surgically treated before any study procedure.
* Existence of bacterial, fungal or viral infections severe or uncontrolled that, in the opinion of the principal investigator, could interfere with the patient's participation in the study or the assessments of the study results.
* Any illness or medical condition that is unstable or can put patient safety at risk and compliance in the study.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: ART patients, with indication of diagnosis of endometrial receptivity by ERA that will receive embryo transfer with frozen blastocyst stage embryos (day 5/day 6).
Sampling Method: Non-Probability Sample
Enrollment: 452 (Actual)
Dates: Start 2017-08-04 (Actual); Primary Completion 2019-05-17 (Actual); Study Completion 2020-06-25 (Actual)

PRIMARY OUTCOMES:
Development of a new non-invasive diagnosis test of Endometrial Microbiome (EM) in infertile patients | 24 months
  Bacterial DNA analysis by Next Generation Sequencing (NGS) using endometrial fluid for the EM diagnose. This will be measured by the percentage of each bacterial DNA in EF samples

SECONDARY OUTCOMES:
Live birth rate | 40 weeks
  Number of babies born per embryo transfer
Implantation rate | 12 weeks
  Number of implanted embryos per total number of embryos transferred
Pregnancy rate | 20 weeks
  Number of pregnancies per embryo transfer
Biochemical pregnancies | 20 weeks
  Number of biochemical pregnancies per total number of pregnancies
Ectopic pregnancies | 20 weeks
  Number of ectopic pregnancies per total number of pregnancies
Clinical miscarriages | 20 weeks
  Number of clinical miscarriages per total number of pregnancies
Ongoing pregnacy rate | 40 weeks
  Number of ongoing pregnancies per embryo transfer

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Simón, MD PhD, Study Chair — Igenomix
Locations (13):
- United States (4):
  - RMA Connecticut, Norwalk, Connecticut
  - IVF Florida, Margate, Florida
  - Missouri Center for Reproductive Medicine (MCRM Fertility), Chesterfield, Missouri
  - Dominion Fertility, Arlington, Washington
- Argentina (2):
  - Gestanza Medicina Reproductiva, Rosario, Santa Fe Province
  - Pregna Medicina Reproductiva, Buenos Aires
- Pacific Center for Reproductive Medicine, Burnaby, British Columbia, Canada
- oak Clinic Sumiyoshi, Osaka, Osaka, Japan
- Alpha Fertility Center, Petaling Jaya, Selangor, Malaysia
- New Hope Fertility Center, Mexico City, Mexico
- Spain (2):
  - Clinica Fertia, Fuengirola, Malaga
  - ProcreaTec, Madrid
- Bahçeci Fulya IVF Center, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No